CLINICAL TRIAL: NCT02777957
Title: Predictors and Survival in Pulmonary Hypertension Associated With Severe Lung Disease
Brief Title: Predictors of Pulmonary Hypertension in Patients With Advanced Lung Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Silesian Centre for Heart Diseases (Other)
Responsible Party: Principal Investigator, Jolanta Nowak, MD, PhD, Silesian Centre for Heart Diseases
Other Study IDs: SilesianCHD
Record Dates: First submitted 2016-05-18; First posted 2016-05-19 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Hypertension
Keywords: Echocardiography; Lung Transplantation
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- mPAP ≥ 25 mmHg: mean pulmonary artery pressure (mPAP) ≥ 25 mmHg (37 patients)
- mPAP < 25 mmHg: mean pulmonary artery pressure (mPAP) < 25 mmHg (28 patients).

SUMMARY:
First, the aim of the study was to evaluate the usefulness of echocardiographic parameters for detecting pulmonary hypertension (PH) in patients with advanced lung disease referred for lung transplantation. Second, to assess the prevalence of PH and to identify which hemodynamic, echocardiographic, pulmonary functional test, exercise capacity and biochemical parameters (especially NT-proBNP) have an impact on survival in a cohort of patients with severe lung diseases referred for lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* advanced lung disease
* qualification for lung transplantation
* written informed consent
* pulmonary capillary wedge pressure < 15 mmHg

Exclusion Criteria:

* cancer,
* history of idiopathic pulmonary hypertension,
* primary valvular heart diseases,
* coronary artery disease,
* collagen vascular disease,
* history or evidence of left ventricular dysfunction,
* atrial fibrillation,
* increased liver enzyme levels ( 3 times the upper laboratory limit),
* renal dysfunction (estimated glomerular filtration rate < 60 ml/min/1.73m2)
* patients who didn't write the personal informed consent
* any specific therapy for PH.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with advanced lung diseases referred for lung transplantation. All patients underwent examinations as potential candidates for lung transplantation, including laboratory testing, pulmonary function tests, exercise capacity, echocardiography examination, and right heart catheterization. Evaluation for lung transplantation was performed during clinically stable periods in all patients on optimal medical and oxygen therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-12; Primary Completion 2020-04 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Survival after the initial right heart catheterization (RHC) measurements | 1 year

SECONDARY OUTCOMES:
Survival to lung transplantation or the end of the observation period after the initial right heart catheterization (RHC) measurement | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Nowak, MD, PhD, Principal Investigator — 3rd Department of Cardiology, Silesian Centre for Heart Diseases; Mariusz Gasior, Prof., PhD, Study Chair — 3rd Department of Cardiology, Silesian Centre for Heart Diseases; Slawomir Zeglen, MD, PhD, Study Chair — Departament of Cardiac Surgery and Transplantology, Silesian Centre for Heart Diseases; Jacek Wojarski, MD, PhD, Study Chair — Departament of Cardiac Surgery and Transplantology, Silesian Centre for Heart Diseases
Locations (1):
- Silesian Centre for Heart Diseases, Zabrze, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nowak J, Hudzik B, Jastrzebski D, Niedziela JT, Rozentryt P, Wojarski J, Ochman M, Karolak W, Zeglen S, Gierlotka M, Gasior M. Pulmonary hypertension in advanced lung diseases: Echocardiography as an important part of patient evaluation for lung transplantation. Clin Respir J. 2018 Mar;12(3):930-938. doi: 10.1111/crj.12608. Epub 2017 Jan 12. PMID 28052583